CLINICAL TRIAL: NCT00280943
Title: Secondary Prevention of Osteoporotic Fractures in Residents of Long-Term Care Facilities Written for FDA Approved Medications for Osteoporosis Treatment.
Brief Title: Secondary Prevention of Osteoporotic Fractures in Residents of Long-Term Care Facilities
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 4686-05-7R2ER
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2007-10

CONDITIONS: Hip Fractures; Osteoporosis
Keywords: All NC LTC facilities having ten residents with a hip fracture or osteoporosis on the MDS will be invited to participate in the trial
MeSH Terms: conditions — Hip Fractures; Osteoporosis | interventions — Home Nursing

INTERVENTIONS:
Behavioral: Long-term care facilities in the intervention arm will receive education and feedback audit on performance

SUMMARY:
Osteoporotic fractures of the hip are a major cause of admission to long-term care facilities. Such fractures put patients at high risk for further fractures, pain and disability. Current data show that many patients in long-term care facilities do not receive FDA medications for their osteoporosis. This trial will test whether a multi-model intervention (which provides feedback about provider use of osteoporosis medications, information about osteoporosis, and currently approved osteoporosis medications)directed at physicians, other health care providers, and nurses will improve the number of prescriptions written for FDA approved medications for osteoporosis treatment.

ELIGIBILITY:
Inclusion Criteria:

Any North Carolina long-term care facility with ten residents who had had a hip fracture or osteoporosis diagnosis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 2005-01; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Number of new prescriptions for FDA-Approved osteoporosis medications.

SECONDARY OUTCOMES:
Secondary Outcome Measures: Changes in number of bone mineral density test ordered, change in the number of hip protectors issued, change in the number of prescriptions for calcium and vitamin D, changes in the rate of new osteoporotic fractures.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth W Lyles, M.D., Principal Investigator — Duke University; Cathleen S. Colon-Emeric, MD, MHSc, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Colon-Emeric CS, Lyles KW, House P, Levine DA, Schenck AP, Allison J, Gorospe J, Fermazin M, Oliver K, Curtis JR, Weissman N, Xie A, Saag KG. Randomized trial to improve fracture prevention in nursing home residents. Am J Med. 2007 Oct;120(10):886-92. doi: 10.1016/j.amjmed.2007.04.020. PMID 17904460